CLINICAL TRIAL: NCT03321890
Title: A Multicenter, Single-arm, Open II Phase Clinical Trial Evaluating the Efficacy of Chidamide Combined With Prednisone, Cyclophosphamide, Etoposide, and Methotrexate (PECM) in Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Brief Title: Chidamide Combined With PECM in Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhiming, Principal Investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-FXY-079-内科
Record Dates: First submitted 2017-02-18; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: relapsed or refractory; peripheral T-cell lymphoma; Combination therapy
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Recurrence | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Prednisone; Cyclophosphamide; Etoposide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination therapy regimen (Experimental): Chidamide + prednisone+cyclophosphamide+etoposide+methotrexate
  Interventions: Drug: Chidamide; Drug: prednisone; Drug: Cyclophosphamide; Drug: etoposide; Drug: Methotrexate

INTERVENTIONS:
Drug: Chidamide — Oral, each taking 30 mg (6 tablets), medication twice a week, 30 minutes after breakfast
Drug: prednisone — oral, 20mg / day,after breakfast
Drug: Cyclophosphamide — oral, 50mg / day,after lunch
Drug: etoposide — oral, 50mg / day,after dinner
Drug: Methotrexate — oral, 10mg / times, once a week,after breakfast

SUMMARY:
To observe the efficacy and safety of Chidamide combined with prednisone, cyclophosphamide, etoposide and methotrexate in relapsed or refractory PTCL.

DETAILED DESCRIPTION:
Prednisone, cyclophosphamide, etoposide, and methotrexate regimens are derived from a "metronidazole, etoposide, procarbazine and cyclophosphamide (PEPC) regimen" regimen that differs from the traditional "maximal Tolerance "chemotherapy, and the use of low-dose chemotherapy, frequent drug therapy, the purpose is to anti-angiogenesis and reduce drug resistance. At present, the program in our treatment of relapsed or refractory PTCL patients effective, safe and controllable, but also look forward to other joint treatment, so as to achieve better curative effect. To provide new treatment options for such patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed peripheral T-cell lymphoma (PTCL) patients;
2. Patients who have had at least one systemic treatment (including chemotherapy, hematopoietic stem cell transplantation, etc.) who have not remission or relapsed after remission;
3. For various reasons can not be hematopoietic stem cell transplantation in patients;
4. The age of 18-75 years old, male, female open;
5. ECOG (Eastern Cooperative Oncology Group) physical scoring 0-1 points;
6. Absolute value of neutrophil≥1.5 × 109 / L, platelet≥90 × 109 / L, hemoglobin≥90g / L;
7. The expected survival time ≥ 3 months;
8. No radiotherapy, chemotherapy, targeted therapy or hematopoietic stem cell transplantation were performed within 4 weeks prior to enrollment.
9. Voluntary signature of written informed consent.

Exclusion Criteria:

1. Pregnancy, breastfeeding women and unwilling to take contraceptive measures of reproductive age patients;
2. B-mode ultrasonography showed that the width of end-diastolic pericardial dark area was ≥10mm;
3. Patients receiving organ transplants;
4. Patients receiving symptomatic treatment of pre-bone marrow toxicity within 7 days prior to enrollment;
5. Patients with active bleeding;
6. Liver function abnormalities (total bilirubin> 1.5 times the upper limit of normal, ALT( alanine aminotransferase) / AST (Aspartate aminotransferase)> 2.5 times the upper limit of normal or hepatic involvement of ALT / AST> 5 times the upper limit of normal), renal dysfunction Creatinine> 1.5 times the upper limit of normal), electrolyte abnormalities;
7. Persons with mental disabilities / those who can not obtain informed consent;
8. Patients with drug abuse and long-term alcohol abuse that may affect the evaluation of test results;
9. The investigators determined that they were not fit to participate in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2017-03-07 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | every 8 weeks until 2 years after last patient's enrollment
  the total proportion of patients with complete response（CR or CRu）and partial response（PR）

SECONDARY OUTCOMES:
Duration of response | every 8 weeks until 2 years after last patient's enrollment
  Duration of complete response（CR or CRu）and partial response（PR）
Progress Free Survival(PFS) | 2 years
  Time from treatment until disease progression or death
Overall Survival | 2 years
  Time from treatment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Wenqi Jiang, MD, Principal Investigator — Department of Medical Oncology,Sun Yat-Sen University
Locations (1):
- Department of Medical Oncology,Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided